CLINICAL TRIAL: NCT04947761
Title: Modified Tian Wang Bu Xin Dan Hydrogel Patch in Preventing Postoperative Delirium in Elderly Patients: A Muticenter Randomised Control Trial
Brief Title: Modified Tian Wang Bu Xin Dan Hydrogel Patch in Preventing Postoperative Delirium in Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TWBXDPOD
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Cheonwangbosimdan Hydrogel patch (Experimental): Group receiving modified Cheonwangbosimdan Hydrogel patch
  Interventions: Drug: modified Tian Wang Bu Xin Dan hydrogel patch
- Placebo patch (Placebo Comparator): Group receiving placebo patch
  Interventions: Other: placebo patch

INTERVENTIONS:
Drug: modified Tian Wang Bu Xin Dan hydrogel patch — modified Cheonwangbosimdan hydrogel patch (one patch/24 hours) applied to Shenque point for 4 days (1 patch daily beginning 2 days preoperative, and continued at 1 patch daily until 2 days postoperatively)
  Other Names: modified Cheonwangbosimdan hydrogel patch
  Arms: modified Cheonwangbosimdan Hydrogel patch
Other: placebo patch — placebo patch (one patch/24 hours) applied to Shenque point for 4 days (1 patch daily beginning 2 days preoperative, and continued at 1 patch daily until 2 days postoperatively)
  Arms: Placebo patch

SUMMARY:
The purpose of this study is to determine whether preoperative administration of Modified Tian Wang Bu Xin Dan Hydrogel Patch prevents the incidence of postoperative delirium in elderly patients undergoing major surgery.

DETAILED DESCRIPTION:
The Traditional Chinese Medicine (TCM) Tian Wang Bu Xin Dan (TWBXD, Cheonwangbosimdan), first recorded in Effective Formulae Handed Down for Generations ( Shi Yi De Xiao Fang) in 1337, is a herbal medicine that has been continuously utilized in Chinese medicine. It alleviates insomnia, anxiety, and palpitation by furnishing energy and stabilizing patients' mind. Cheonwangbosimdan can mitigate primary insomnia and secondary insomnia in patients with hyperthyroidism and menopause without severe side effects.

Tianwang Buxin Decoction has the same effect as Olanzapine for the treatment of delirium after hip joint replacement in falling-induced senile femoral neck fracture patients.

This study aim to evaluate the incidence of postoperative delirium in elderly patients treated with prophylactic Modified Cheonwangbosimdan Hydrogel Patch versus placebo patch.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥70 years;
2. Underwent elective non-cardiac surgery (including Orthopedics, thoracic, urology, general surgery patients)under general anesthesia ;

Exclusion Criteria:

1. History of neuropsychiatric diseases including delirium, mental disorders, Parkinson, dementia, etc.;
2. The operation was cancelled due to various reasons after the patient was enrolled;
3. severe liver disease; severe renal dysfunction defined as either having creatinine clearance < 30 ml/min or being dialysis-dependent;
4. Patients who undergo second operation in a short period;
5. Past 30-day prescribed use of sedative-hypnotics for the indication of insomnia;
6. History of alcohol abuse or a history of drug dependence;
7. Cannot with the completion of tests of cognitive function;
8. Known allergy to skin patch;
9. Treatment site has active skin lesion or inflammation;
10. Refused to participate in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of inpatient post-operative delirium as measured using the 3D-confusion assessment method (3D-CAM) | Day 1 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of inpatient post-operative delirium as measured using the 3D-confusion assessment method (3D-CAM) | Day 2 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of inpatient post-operative delirium as measured using the 3D-confusion assessment method (3D-CAM) | Day 3 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily

SECONDARY OUTCOMES:
Sleep Quality | Baseline and 1,3 days after surgery
  Objective sleep quality will be measured using a Fitbit Charge 3 activity monitor to be worn
Athens Insomnia Scale | Baseline and 1,2,3 days after surgery
  using the Athens Insomnia Scale to test the subjective sleep quality of patients. The range were from 0-3. Total score < 4 means sleep well; total score =6 means suspicious of insomnia; total score > 6 means insomnia.
Pain at rest using Numerical Rating Scale(NRS) | postoperative days 1, 2, 3
  NRS pain scores will also be measured at rest. The NRS is a validated 11-point numerical scale that ranges from 0 (no pain) to 10 (worst pain possible).
Total postoperative analgesic requirements | First 48 hours postoperatively
  Amount of opioid (IV morphine or hydromorphone) and oral analgesics required for pain control, reported as overall morphine equivalents.
Change in biological markers (1) | Baseline and 1 day after surgery
  Plasma levels of CXCL13
Change in biological markers (2) | Baseline and 1 day after surgery
  Plasma levels of S100B
STOP-Bang score | Baseline
  STOP-BANG questionnaire
Pittsburgh Sleep Quality Index | Baseline and day 3 postoperatively
  The PSQI is filled out by the patient and assesses patient sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Director — Chinese PLA General Hospital
Locations (3):
- China (3):
  - Fifth Medical center of Chinese PLA General Hospital, Beijing
  - First Medical center of Chinese PLA General Hospital, Beijing
  - Fourth Medical center of Chinese PLA General Hospital, Beijing